CLINICAL TRIAL: NCT03056911
Title: Clinical Effects of Ozone Therapy in Cervical Disc Hernia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, Assistant Professor, Sakarya University
Other Study IDs: sakarya Ozone
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Pain, Neck
Keywords: ozone therapy; percutaneous treatment; Oswestry Disability Index (ODI); Visual analog Scale (VAS); Neuropathic Pain Questionnaire (DN-4); cervical
MeSH Terms: conditions — Neck Pain | interventions — Ozone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ozone: Chemonucleolysis by ozone therapy Patients visiting the pain clinic of the hospital who had cervical discogenic or radicular pain that did not resolve after the use of conventional therapy. Written informed consent was obtained from all participants.
  Interventions: Drug: Ozone

INTERVENTIONS:
Drug: Ozone — Pain relief with chemonucleolysis by using ozone regard to age, sex, ASA score, and complications.

SUMMARY:
The aim of the study is to evaluate the clinical effects of Ozone-oxygen therapy as therapeutic substance for nucleolysis application in the patients with cervical disc hernia who had chronic pain and weakness on the neck, shoulders and arms

DETAILED DESCRIPTION:
This is a retrospective, single-center study that is going to be conducted from November 2013 to May 2016 on patients visiting the pain clinic of the hospital who were treated with Ozone-oxygen therapy for cervical discogenic or radicular pain.

Data collected from medical record forms and electronic medical record system of the hospital were used in the retrospective analysis of medical data with regard to age, gender, complications.

A resident who has not involved in the study interviewed each patient by telephone on the follow up to collect the related information.

ELIGIBILITY:
Inclusion Criteria:

* continuous radicular pain radiating to the upper limb, with a duration ≥8 weeks and an intensity >4/10 as rated by the patient on a visual analog scale (VAS)
* resistant to appropriate conservative treatment combining antiinflammatory drugs, and confirmed by imaging with CT or MRI of a herniated disc putting pressure on a nerve root consistent with the clinical pain.

Exclusion Criteria:

* history of surgery at the cervical spine, contraindication to percutaneous chemonucleolysis (coagulopathy or infection), imaging results that did not support the clinical results, the presence of a herniated disc excluded or calcified on imaging, possible interference with pain evaluation due to any medical condition or treatment, involvement of incomplete data collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted from November 2013 to May 2016 on patients visiting the pain clinic who had cervical diskogenic or radicular pain that did not resolve after the use of conventional therapy.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score for pain | 1 month
  Ozone therapy technique for pain relief assessed by Statistical Package for the Social Sciences (SPSS) v22.0 Statistical assessment of each patient was evaluated on time intervals before procedure, in the 1st month after procedure for Visual analogue scale (VAS) score for pain

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) score | 3 months
  Assessment of degree of disability and estimating quality of life based on Oswestry Disability Index (ODI) score by SPSS v22.0 Statistical assessment of each patient was evaluated on time intervals before procedure, in the 3rd months after procedure for ODI score
ODI score | 1 month
  Assessment of degree of disability and estimating quality of life based on Oswestry Disability Index (ODI) score by SPSS v22.0 Statistical assessment of each patient was evaluated on time intervals before procedure, in the 1st month after procedure for ODI score

CONTACTS AND LOCATIONS:
Overall Officials: Serbülent Beyaz, AssocProf, Study Chair — Sakarya University Research and Training Hospital
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Magalhaes FN, Dotta L, Sasse A, Teixera MJ, Fonoff ET. Ozone therapy as a treatment for low back pain secondary to herniated disc: a systematic review and meta-analysis of randomized controlled trials. Pain Physician. 2012 Mar-Apr;15(2):E115-29. PMID 22430658